CLINICAL TRIAL: NCT03642223
Title: Relation Btw Adiposity, Inflammation & Iron Absorption:Comparison Btw Central & Peripheral Adiposity
Brief Title: Central and Peripheral Adiposity and Iron Absorption
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swiss Federal Institute of Technology (Other)
Collaborators: American University of Beirut Medical Center (Other)
Responsible Party: Principal Investigator, Prof. Michael B. Zimmermann, Prof. Dr. med., Swiss Federal Institute of Technology
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: FLAB
Record Dates: First submitted 2018-07-24; First posted 2018-08-22 (Actual); Last update posted 2019-03-28 (Actual); Status verified 2019-03

CONDITIONS: Adiposity; Iron-deficiency
MeSH Terms: conditions — Obesity; Anemia, Iron-Deficiency

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- normal-weight (Active Comparator)
  Interventions: Other: Stable iron isotopes
- peripheral adiposity (Experimental)
  Interventions: Other: Stable iron isotopes
- central adiposity (Experimental)
  Interventions: Other: Stable iron isotopes

INTERVENTIONS:
Other: Stable iron isotopes — Participants have to consume a test meal containing stable iron isotopes in order to determine iron absorption

SUMMARY:
Adiposity is a state of sub-clinical inflammation, thus hepcidin is increased in adiposity, often leading to iron deficiency in this population group. Central adiposity is generally considered having a greater negative effect on health compared to peripheral adiposity. Whether this can be also seen in hepcidin and thereby in iron absorption is uncertain.

ELIGIBILITY:
Inclusion Criteria:

* either normal-weight (BMI 18-25kg/m2) or overweight/obese (BMI 28-50kg/m2) with either central or peripheral fat deposits based on DEXA

Exclusion Criteria:

* Iron Supplement or antibiotic intake within 2 weeks before study start
* diagnosed chronic disease or gastrointestinal disorders
* regular use of medication (except contraceptives)
* pregnancy
* lactation
* smoking
* blood donation or surgery within the last 4 months.

Ages: 20 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 121 (Actual)
Dates: Start 2017-09-10 (Actual); Primary Completion 2018-10-18 (Actual); Study Completion 2018-10-18 (Actual)

PRIMARY OUTCOMES:
Fractional and total iron absorption | 14days after the administration of the test meal

SECONDARY OUTCOMES:
Serum Hepcidin | at baseline
Serum ferritin | at baseline
  iron status
Serum TfR | at baseline
  iron status
Serum CRP | at baseline
  inflammation status
Serum AGP | at baseline
  inflammation status
Serum IL-6 | at baseline
  inflammation status

CONTACTS AND LOCATIONS:
Locations (1):
- American University of Beirut, Beirut, Lebanon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] El-Helou N, El-Mallah C, Wehbe N, Bissani N, Stoffel N, Herter-Aeberli I, Zimmermann M, Obeid O. A test to measure oral iron absorption and glucose tolerance simultaneously in 18 to 55 year old premenopausal women. Clin Nutr ESPEN. 2021 Dec;46:325-329. doi: 10.1016/j.clnesp.2021.09.737. Epub 2021 Sep 29. PMID 34857214